CLINICAL TRIAL: NCT06206668
Title: Effect of Referent Type on Balance in Action Observation in Healthy People: Randomized Clinical Trial.
Brief Title: Effect of Referent Type on Balance in Action Observation.
Acronym: ROA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Tania López Hernández, Principal Investigator, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01/2023
Record Dates: First submitted 2023-12-31; First posted 2024-01-16 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Balance Disorders
Keywords: Action observation; Referent; Gender; Balance
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Participants will watch a video of landscapes without human or animal movement.
- Intervention Group with Referent (GIR) (Experimental): Participants will observe actions whose referent has been selected by themselves based on perceived similarity. A total of 16 different videos will be used, with 4 new videos each week. The videos will gradually increase in difficulty as the study progresses. All exercises are exercises used to improve balance.
  Interventions: Other: Action observation videos
- Standard Intervention Group (GIE) (Active Comparator): Participants will observe actions with a standard reference. In this case, a basic digitally designed faceless doll will be used. A total of 16 different videos will be used, with 4 new videos each week. The videos will gradually increase in difficulty as the study progresses. All exercises are exercises used to improve balance.
  Interventions: Other: Action observation videos

INTERVENTIONS:
Other: Action observation videos — The participant will see videos of balance exercises performed by the assigned reference, depending on their group, without performing any physical movement.
  Arms: Intervention Group with Referent (GIR); Standard Intervention Group (GIE)

SUMMARY:
The objective of the study is to analyze whether observing the actions of a referent selected by the participants improves balance in asymptomatic individuals compared to those who observe a standard referent.

DETAILED DESCRIPTION:
Design: Randomized controlled clinical trial. The primary endpoint of the study was the balance recorded by force platform (estatic) and Y balance test (dynamic).

Setting: The participants will be healthy people in the province of Tarragona.

Participants: They will be randomly assigned to one of three groups using a computerized randomized list:

* Control Group (CG): Participants will watch a video of landscapes without human or animal movement.
* Intervention Group with Referent (GIR): Participants will observe actions whose referent has been selected by themselves based on perceived similarity.
* Standard Intervention Group (GIE): Participants will observe actions with a standard reference.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age.
* Have a mobile device.
* Have normal or corrected-to-normal vision.
* Absence of neurological, orthopedic or vestibular disorders.
* Absence of specific balance skills due to competitive sports.
* Obtain a score of 3 or less on the Tegner activity scale.
* Having voluntarily signed the informed consent and being willing to follow the protocol proposed by the research team.

Exclusion Criteria:

* History of participation in any study with movement representation methods.
* Subjects with impaired communication and/or compression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Static balance | 1 month
  Center of pressure analysis: The displacement of the center of pressure (CPD) of the participants will be measured through posturographic tests performed on a force platform. The following variables related to the center of pressure (CoP) will be calculated: the roll area (in square millimeters) and the distribution of the weight load on both sides.
Dynamic Balance | 1 month
  A modified and abbreviated version of the Star Excursion Balance Test, known as mSEBT, will be used. This test has been standardized and validated, and requires a board or floor with three lines indicating directions of movement: anterior (ANT), posteromedial (PM), and posterolateral (PL). These lines form a Y, with an angle of 90° between PM and PL, and 135° between ANT and PM, and ANT and PL.

SECONDARY OUTCOMES:
Age | 1 day
  Age will be measured in years
Biological sex | 1 day
  Biological sex will be measured asking if they born like a boy or a girl.
Weight | 1 day
  Weight will be measured in kg with a Beurer's body analyser scales
Height | 1 day
  Height will be measured in cm.
Body mass index (BMI) | 1 day
  Body mass index (BMI) will be measured in kg with a Beurer's body analyser scales
Length of the lower limb. | 1 day
  Length of the lower limb will be measured in cm.
Dominant lower limb | 1 day
  Dominant lower limb will be measured asking which limb would shoot a ball with.
Morphotype | 1 day
  Morphotype (endomorph, ectomorph and mesoform) will be measured by observation
Trunk and lower extremity muscle strength | 1 month
  Analogue dynamometry will be used as an evaluation method and will be recorded in Newtons (N) with the Saehan SKU SH5007 back, leg and chest dynamometer.
Satisfaction assessed by a selfcreate questionnaire | 1 day
  A questionnaire specifically designed to evaluate participants' satisfaction with their experience in the study will be used once they have completed their participation.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Adillón Camón, Dra., Study Director — University Rovira i Virgili
Locations (1):
- Centre Tecnològic de Nutrició i Salut Eurecat, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gatti R, Sarasso E, Pelachin M, Agosta F, Filippi M, Tettamanti A. Can action observation modulate balance performance in healthy subjects? Arch Physiother. 2019 Jan 22;9:1. doi: 10.1186/s40945-018-0053-0. eCollection 2019. PMID 30693101
- [Background] Moon Y, Bae Y. The effect of backward walking observational training on gait parameters and balance in chronic stroke: randomized controlled study. Eur J Phys Rehabil Med. 2022 Feb;58(1):9-15. doi: 10.23736/S1973-9087.21.06869-6. Epub 2021 Sep 1. PMID 34468110
- [Background] Picot B, Terrier R, Forestier N, Fourchet F, O.McKeon F. The Star Excursion Balance Test: An Update Review and Practical Guidelines. Int. J. Athl. Ther. Train. 2021 Jul 20,26(6):285-93. doi: 10.1123/ijatt.2020-0106.
- [Background] Leem SH, Kim JH, Lee BH. Effects of Otago exercise combined with action observation training on balance and gait in the old people. J Exerc Rehabil. 2019 Dec 31;15(6):848-854. doi: 10.12965/jer.1938720.360. eCollection 2019 Dec. PMID 31938708
- [Background] Cuenca-Martinez F, Suso-Marti L, Sanchez-Martin D, Soria-Soria C, Serrano-Santos J, Paris-Alemany A, La Touche R, Leon-Hernandez JV. Effects of Motor Imagery and Action Observation on Lumbo-pelvic Motor Control, Trunk Muscles Strength and Level of Perceived Fatigue: A Randomized Controlled Trial. Res Q Exerc Sport. 2020 Mar;91(1):34-46. doi: 10.1080/02701367.2019.1645941. Epub 2019 Oct 18. PMID 31626568